CLINICAL TRIAL: NCT02200614
Title: A Multinational, Randomised, Double-blind, Placebo-controlled, Phase III Efficacy and Safety Study of Darolutamide (ODM-201) in Men With High-risk Non-metastatic Castration-resistant Prostate Cancer
Brief Title: Efficacy and Safety Study of Darolutamide (ODM-201) in Men With High-risk Non-metastatic Castration-resistant Prostate Cancer
Acronym: ARAMIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17712; 2013-003820-36 (EudraCT Number)
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer Non-Metastatic; Castration-Resistant
MeSH Terms: interventions — darolutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Darolutamide (BAY1841788) (Experimental): Participants received Darolutamide 600 mg (2 tablets of 300 mg) twice daily with food, equal to a total daily dose of 1200 mg.
  Interventions: Drug: Darolutamide (Nubeqa, BAY1841788)
- Placebo (Placebo Comparator): Participants received matching placebo 2 tablets twice daily with food.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darolutamide (Nubeqa, BAY1841788) — Darolutamide 600 mg (2 tablets of 300 mg) twice daily with food, equivalent to a total daily dose of 1200 mg.
  Other Names: ODM-201
  Arms: Darolutamide (BAY1841788)
Drug: Placebo — Matching placebo 2 tablets twice daily with food.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of BAY1841788 (ODM-201) in patients with non-metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of prostate without neuroendocrine differentiation or small cell features.
* Castration-resistant prostate cancer (CRPC) with castrate level of serum testosterone.
* Prostate-specific Antigen (PSA) doubling time of ≤ 10 months and PSA > 2ng/ml.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Blood counts at screening: haemoglobin ≥ 9.0 g/dl,absolute neutrophil count ≥ 1500/µl, platelet count ≥ 100,000/µl.
* Screening values of serum alanine aminotransferase (ALT) and/or aspartate transaminase (AST) ≤ 2.5 x upper limit of normal (ULN), total bilirubin ≤ 1.5 x ULN, creatinine ≤ 2.0 x ULN.
* Sexually active patients, unless surgically sterile, must agree to use condoms as an effective barrier method and refrain from sperm donation during the study treatment and for 3 months after the end of the study treatment.

Exclusion Criteria:

* History of metastatic disease at any time or presence of detectable metastases.
* Acute toxicities of prior treatments and procedures not resolved to grade ≤ 1 or baseline before randomisation.
* Prior treatment with: second generation androgen receptor (AR) inhibitors, other investigational AR inhibitors, or CYP17 enzyme inhibitor.
* Use of estrogens or 5-α reductase inhibitors or AR inhibitors.
* Prior chemotherapy or immunotherapy for prostate cancer.
* Use of systemic corticosteroid.
* Radiation therapy within 12 weeks before randomisation.
* Severe or uncontrolled concurrent disease, infection or co-morbidity.
* Treatment with bisphosphonate or denosumab within 12 weeks before randomisation.
* Known hypersensitivity to the study treatment or any of its ingredients.
* Major surgery within 28 days before randomisation.
* Any of the following within 6 months before randomisation: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft; congestive heart failure New York Heart Association (NYHA) Class III or IV.
* Uncontrolled hypertension.
* Prior malignancy.
* Gastrointestinal disorder or procedure which expects to interfere significantly with absorption of study treatment.
* Active viral hepatitis, active human immunodeficiency virus (HIV) or chronic liver disease.
* Treatment with any investigational drug within 28 days before randomisation.
* Any condition that in the opinion of the investigator would impair the patients' ability to comply with the study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1509 (Actual)
Dates: Start 2014-09-12 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2021-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (338):
- United States (51):
  - Homewood, Alabama
  - Anchorage, Alaska
  - Tucson, Arizona
  - Fountain Valley, California
  - La Jolla, California
  - Laguna Hills, California
  - Los Angeles, California
  - San Diego, California
  - Whittier, California
  - Denver, Colorado
  - Parker, Colorado
  - Boca Raton, Florida
  - Orlando, Florida
  - Port Saint Lucie, Florida
  - Coeur d'Alene, Idaho
  - Chicago, Illinois
  - Evanston, Illinois
  - Springfield, Illinois
  - Greenwood, Indiana
  - Indianapolis, Indiana
  - Jeffersonville, Indiana
  - West Des Moines, Iowa
  - Wichita, Kansas
  - New Orleans, Louisiana
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Salisbury, Maryland
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - Royal Oak, Michigan
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Voorhees Township, New Jersey
  - Syracuse, New York
  - The Bronx, New York
  - Asheboro, North Carolina
  - Charlotte, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Gahanna, Ohio
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Bala-Cynwyd, Pennsylvania
  - Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Fairfax, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Wheeling, West Virginia
- Argentina (5):
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Santa Fé, Santa Fe Province
  - San Miguel de Tucumán, Tucumán Province
  - Córdoba
  - La Rioja
- Australia (6):
  - Randwick, New South Wales
  - St Leonards, New South Wales
  - Douglas, Queensland
  - South Brisbane, Queensland
  - Kurralta Park, South Australia
  - Fitzroy, Victoria
- Vienna, Austria
- Belarus (2):
  - Lesnoy
  - Minsk
- Belgium (5):
  - Bonheiden
  - Kortrijk
  - Libramont
  - Liège
  - Sint-Truiden
- Brazil (16):
  - Fortaleza, Ceará
  - Salvador, Estado de Bahia
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Juiz de Fora, Minas Gerais
  - Uberlândia, Minas Gerais
  - Curitiba, Paraná
  - Recife, Pernambuco
  - Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Itajaí, Santa Catarina
  - Barretos, São Paulo
  - Jaú, São Paulo
  - Ribeirao Preto - SP, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo
- Bulgaria (2):
  - Sofia
  - Varna
- Canada (9):
  - Calgary, Alberta
  - Halifax, Nova Scotia
  - Burlington, Ontario
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Granby, Quebec
  - Pointe-Claire, Quebec
- Colombia (3):
  - Medellín, Antioquia
  - Montería, Departamento de Córdoba
  - Floridablanca, Santander Department
- Czechia (5):
  - Jablonec nad Nisou
  - Kolín
  - Olomouc
  - Opava
  - Prague
- Tallinn, Estonia
- Finland (5):
  - Helsinki
  - Kuopio
  - Seinäjoki
  - Tampere
  - Turku
- France (25):
  - Angers
  - Bayonne
  - Besançon
  - Bordeaux
  - Caen
  - Cergy-Pontoise
  - Clermont-Ferrand
  - Créteil
  - Dijon
  - La Roche-sur-Yon
  - Limoges
  - Montpellier
  - Nancy
  - Nantes
  - Paris
  - Pierre-Bénite
  - Poitiers
  - Reims
  - Rennes
  - Rouen
  - Saint-Mandé
  - Strasbourg
  - Suresnes
  - Tours
  - Villejuif
- Germany (22):
  - Emmendingen, Baden-Wurttemberg
  - Kirchheim unter Teck, Baden-Wurttemberg
  - Mühlacker, Baden-Wurttemberg
  - Nürtingen, Baden-Wurttemberg
  - Reutlingen, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Zirndorf, Bavaria
  - Frankfurt am Main, Hesse
  - Marburg, Hesse
  - Herzberg am Harz, Lower Saxony
  - Holzminden, Lower Saxony
  - Hagenow, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Mülheim, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Magdeburg, Saxony-Anhalt
  - Berlin
  - Hamburg
- Hungary (8):
  - Budapest
  - Debrecen
  - Győr
  - Nyíregyháza
  - Szeged
  - Szekszárd
  - Szolnok
  - Zalaegerszeg
- Haifa, Israel
- Italy (12):
  - Chieti, Abruzzo
  - Lecce, Apulia
  - Catanzaro, Calabria
  - Napoli, Campania
  - Forlì Cesena, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Rome, Lazio
  - Turin, Piedmont
  - Messina, Sicily
  - Palermo, Sicily
  - Arezzo, Tuscany
- Japan (37):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Kurume, Fukuoka
  - Kōriyama, Fukushima
  - Maebashi, Gunma
  - Ōtake, Hiroshima
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Higashiibaraki, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Sendai, Miyagi
  - Ueda, Nagano
  - Kashihara, Nara
  - Yufu, Oita Prefecture
  - Sayama, Osaka
  - Wako, Saitama
  - Hamamatsu, Shizuoka
  - Utsunomiya, Tochigi
  - Bunkyo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Minato-ku, Tokyo
  - Mitaka, Tokyo
  - Nakano-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Sumida-ku, Tokyo
  - Ube, Yamaguchi
  - Chiba
  - Fukui
  - Hiroshima
  - Kyoto
  - Nagasaki
  - Okayama
  - Osaka
  - Toyama
- Latvia (4):
  - Daugavpils
  - Jelgava
  - Leipaja
  - Riga
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Peru (3):
  - La Victoria, Arequipa
  - Lima
  - San Isidro
- Poland (9):
  - Elblag
  - Gdansk
  - Lodz
  - Lublin
  - Otwock
  - Rzeszów
  - Siedlce
  - Warsaw
  - Wroclaw
- Portugal (6):
  - Guimarães, Braga District
  - Almada, Lisbon District
  - Matosinhos Municipality, Porto District
  - Braga
  - Lisbon
  - Porto
- Romania (6):
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Oradea
  - Ploieşti
  - Târgu Mureş
- Russia (17):
  - Chelyabinsk
  - Ivanovo
  - Kazan'
  - Krasnoyarsk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Obninsk
  - Omsk
  - Orenburg
  - Pyatigorsk
  - Rostov-on-Don
  - Saint Petersburg
  - Saratov
  - Tyumen
  - Ufa
  - Vladimir
- Serbia (2):
  - Belgrade
  - Niš
- Slovakia (3):
  - Bratislava
  - Martin
  - Trenčín
- South Africa (6):
  - George, Eastern Cape
  - Port Elizabeth, Eastern Cape
  - Pretoria, Gauteng
  - Paarl, Western Cape
  - Rondebosch, Western Cape
  - Cape Town
- South Korea (6):
  - Gwangju, Gwangju Gwang''yeogsi
  - Cheongju-si, North Chungcheong
  - Seoul, Seoul Teugbyeolsi
  - Daegu
  - Incheon
  - Seoul
- Spain (19):
  - Elche, Alicante
  - Cadiz, Andalusia
  - L'Hospitalet de Llobregat, Barcelona
  - Sabadell, Barcelona
  - Terrassa, Barcelona
  - Jerez de la Frontera, Cádiz
  - Manacor, Illes Baleares
  - Palma de Mallorca, Illes Baleares
  - Alcorcón, Madrid
  - Bilbao, Vizcaya
  - Barcelona
  - Córdoba
  - Granada
  - Lugo
  - Madrid
  - Málaga
  - Salamanca
  - Seville
  - Valencia
- Sweden (4):
  - Gothenburg
  - Örebro
  - Stockholm
  - Uppsala
- Taiwan (5):
  - Kaohsiung City
  - Kaoshiung
  - Taichung
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (5):
  - Ankara
  - Istanbul
  - Izmir
  - Manisa
  - Sivas
- Ukraine (7):
  - Chernivtsi
  - Dnipro
  - Kharkiv
  - Kryvyi Rih
  - Kyiv
  - Uzhhorod
  - Zaporizhzhya
- United Kingdom (17):
  - Reading, Berkshire
  - Llanelli, Carmarthenshire
  - Romford, Essex
  - Stevenage, Hertfordshire
  - Dartford, Kent
  - Maidstone, Kent
  - Preston, Lancashire
  - Bebington, Merseyside
  - Scunthorpe, North East Lincolnshire
  - Bath, Somerset
  - Stoke-on-Trent, Staffordshire
  - Dudley, West Midlands
  - Huddersfield, West Yorkshire
  - Wakefield, West Yorkshire
  - Cardiff
  - Glasgow
  - London

REFERENCES:
- [Derived] Saar M, Fizazi K, Shore ND, Smith M, Damber JE, Semenov A, Ribal MJ, Birtle A, Rigaud J, Wallis CJD, Grimm MO, Halabi S, Armstrong AJ, Mohamed AF, Adorjan P, Srinivasan S, Verholen F, Morgans AK, Siemens DR. Effects of Prior Local Therapy by Radical Prostatectomy or Radiotherapy on the Efficacy and Quality of Life of Patients Treated With Darolutamide in ARAMIS. Cancer Med. 2026 Jan;15(1):e71343. doi: 10.1002/cam4.71343. PMID 41450200
- [Derived] Ni X, Sui J, Wang B, Wang H, Freedland SJ, Ye D, Zhu Y. Lower Testosterone Level and Metastases-Free Survival in Patients With Nonmetastatic Castration-Resistant Prostate Cancer Treated With Novel Antiandrogens: A Post Hoc Analysis of SPARTAN and ARAMIS. J Urol. 2025 Jul;214(1):10-17. doi: 10.1097/JU.0000000000004545. Epub 2025 Mar 25. PMID 40132221
- [Derived] Shore ND, Gratzke C, Feyerabend S, Werbrouck P, Carles J, Vjaters E, Tammela TLJ, Morris D, Aragon-Ching JB, Concepcion RS, Emmenegger U, Fleshner N, Grabbert M, Lietuvietis V, Mahammedi H, Cruz FM, Paula A, Pieczonka C, Rannikko A, Richardet M, Silveira G, Kuss I, Le Berre MA, Verholen F, Sarapohja T, Smith MR, Fizazi K. Extended Safety and Tolerability of Darolutamide for Nonmetastatic Castration-Resistant Prostate Cancer and Adverse Event Time Course in ARAMIS. Oncologist. 2024 Jul 5;29(7):581-588. doi: 10.1093/oncolo/oyae019. PMID 38394384
- [Derived] Fizazi K, Shore ND, Smith M, Ramos R, Jones R, Niegisch G, Vjaters E, Wang Y, Srinivasan S, Sarapohja T, Verholen F. Efficacy and safety outcomes of darolutamide in patients with non-metastatic castration-resistant prostate cancer with comorbidities and concomitant medications from the randomised phase 3 ARAMIS trial. Eur J Cancer. 2023 Oct;192:113258. doi: 10.1016/j.ejca.2023.113258. Epub 2023 Jul 27. PMID 37660438
- [Derived] Carles J, Medina-Lopez RA, Puente J, Gomez-Ferrer A, Nebra JC, Saez Medina MI, Ribal MJ, Antolin AR, Alvarez-Ossorio JL, Suarez Novo JF, Agut CM, Srinivasan S, Ortiz J, Fizazi K. Darolutamide in Spanish patients with nonmetastatic castration-resistant prostate cancer: ARAMIS subgroup analysis. Future Oncol. 2023 Apr;19(12):819-828. doi: 10.2217/fon-2022-1131. Epub 2023 May 24. PMID 37222151
- [Derived] Shore ND, Stenzl A, Pieczonka C, Klaassen Z, Aronson WJ, Karsh L, Ryan CJ, Ortiz J, Srinivasan S, Mohamed AF, Verholen F. Impact of darolutamide on local symptoms: pre-planned and post hoc analyses of the ARAMIS trial. BJU Int. 2023 Apr;131(4):452-460. doi: 10.1111/bju.15887. Epub 2022 Sep 29. PMID 36087070
- [Derived] Chowdhury S, Oudard S, Uemura H, Joniau S, Dearden L, Capone C, Van Sanden S, Diels J, Hadaschik BA. Apalutamide Compared with Darolutamide for the Treatment of Non-metastatic Castration-Resistant Prostate Cancer: Efficacy and Tolerability in a Matching-Adjusted Indirect Comparison. Adv Ther. 2022 Jan;39(1):518-531. doi: 10.1007/s12325-021-01885-6. Epub 2021 Nov 19. PMID 34797506
- [Derived] Fizazi K, Blue I, Nowak JT. Darolutamide and survival in nonmetastatic, castration-resistant prostate cancer: a patient perspective of the ARAMIS trial. Future Oncol. 2021 May;17(14):1699-1707. doi: 10.2217/fon-2020-1291. Epub 2021 Feb 8. PMID 33554636
- [Derived] Fizazi K, Shore N, Tammela TL, Ulys A, Vjaters E, Polyakov S, Jievaltas M, Luz M, Alekseev B, Kuss I, Le Berre MA, Petrenciuc O, Snapir A, Sarapohja T, Smith MR; ARAMIS Investigators. Nonmetastatic, Castration-Resistant Prostate Cancer and Survival with Darolutamide. N Engl J Med. 2020 Sep 10;383(11):1040-1049. doi: 10.1056/NEJMoa2001342. PMID 32905676
- [Derived] Shore N, Zurth C, Fricke R, Gieschen H, Graudenz K, Koskinen M, Ploeger B, Moss J, Prien O, Borghesi G, Petrenciuc O, Tammela TL, Kuss I, Verholen F, Smith MR, Fizazi K. Evaluation of Clinically Relevant Drug-Drug Interactions and Population Pharmacokinetics of Darolutamide in Patients with Nonmetastatic Castration-Resistant Prostate Cancer: Results of Pre-Specified and Post Hoc Analyses of the Phase III ARAMIS Trial. Target Oncol. 2019 Oct;14(5):527-539. doi: 10.1007/s11523-019-00674-0. PMID 31571095
- [Derived] Fizazi K, Shore N, Tammela TL, Ulys A, Vjaters E, Polyakov S, Jievaltas M, Luz M, Alekseev B, Kuss I, Kappeler C, Snapir A, Sarapohja T, Smith MR; ARAMIS Investigators. Darolutamide in Nonmetastatic, Castration-Resistant Prostate Cancer. N Engl J Med. 2019 Mar 28;380(13):1235-1246. doi: 10.1056/NEJMoa1815671. Epub 2019 Feb 14. PMID 30763142
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 36 countries between 12 September 2014 (first participant first visit) and 14 June 2021 (last participant last visit).
Pre-assignment Details: From 2696 participants who signed informed consent, 1187 participants were discontinued from screening. A total of 1509 participants were randomly assigned to either darolutamide arm or placebo arm. The study was unblinded on 30 OCT 2018 and participants in the placebo arm could cross over to open-label darolutamide treatment.
Groups:
- Darolutamide (BAY1841788): Participants received darolutamide 600 mg (2 tablets of 300 mg) twice daily with food, equal to a total daily dose of 1200 mg. Participants in the darolutamide treatment arm were ongoing with open-label darolutamide treatment (darolutamide double-blind [DB] + open-label [OL]).
- Placebo: Participants received matching placebo 2 tablets twice daily with food. Participants from the placebo arm crossed over to receive open-label darolutamide treatment (placebo-darolutamide cross-over [CO]).
Period: Double Blind Treatment
Arm/Group | Darolutamide (BAY1841788) | Placebo
Started (Randomized) | 955 | 554
Completed (Ongoing with treatment) | 591 | 170
Not Completed | 364 | 384
Not completed — Adverse Event | 86 | 48
Not completed — Confirmed metastasis | 120 | 140
Not completed — Judgment of the investigator | 59 | 99
Not completed — Metastasis by local reading | 1 | 3
Not completed — Other reason | 6 | 2
Not completed — Personal reason | 77 | 85
Not completed — Protocol deviation | 14 | 7
Not completed — Not treated | 1 | 0
Period: Open Label
Arm/Group | Darolutamide (BAY1841788) | Placebo
Started | 591 (Not all participants from treatment period entered follow-up) | 170 (Not all participants from treatment period entered follow-up)
Completed (Moving to roll-over study) | 295 | 114
Not Completed | 296 | 56
Not completed — Adverse Event | 41 | 11
Not completed — Confirmed metastasis | 1 | 0
Not completed — Judgment of the investigator | 29 | 2
Not completed — Metastasis by local reading | 138 | 27
Not completed — Other reason | 22 | 4
Not completed — Personal reason | 60 | 8
Not completed — Protocol deviation | 3 | 2
Not completed — Missing | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Darolutamide (BAY1841788) | Placebo | Total
Number analyzed (Participants) | 955 | 554 | 1509
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.9 (7.8) | 73.2 (8.2) | 73.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 955 | 554 | 1509
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asia | 122 | 71 | 193
  Black or African American | 28 | 24 | 52
  White | 760 | 434 | 1194
  Missing | 36 | 19 | 55
  Other | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Metastasis-Free Survival
Description: Metastasis-Free Survival (MFS) is defined as the time from randomisation to evidence of metastasis or death from any cause, whichever occurs first (cut-off date 15 Nov 2019)
Time Frame: From randomization to the time approximately 385 MFS events were observed (approximately 48 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Darolutamide (BAY1841788) | Placebo
Number analyzed (Participants) | 955 | 554
months | 40.37 [34.33 to NA] — NA = value cannot be estimated due to censored data, insufficient number of participants with events | 18.43 [15.51 to 22.34]
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) vs Placebo; Test type: Superiority; p < 0.000001, Log Rank; Hazard Ratio (HR) = 0.413, 95% CI 2-sided [0.341 to 0.500] — Hazard ratio and 95% Confidence Interval (CI) was based on Cox Regression Model, stratified by Prostate-specific antigen doubling time (PSADT) (≤ 6 months vs. > 6 months) and use of osteoclast-targeted therapy (No, Yes)

2. Secondary Outcome: Overall Survival - Primary Analysis
Description: Overall Survival (OS) was defined as the time from randomization to death due to any cause.
Time Frame: From randomization of the first subject to the time approximatively 140 death events were observed (approximately 48 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Darolutamide (BAY1841788) | Placebo
Number analyzed (Participants) | 955 | 554
months | NA [44.45 to NA] — NA = value cannot be estimated due to censored data, insufficient number of participants with events | NA [NA to NA] — NA = value cannot be estimated due to censored data, insufficient number of participants with events
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) vs Placebo; Test type: Superiority; p = 0.045210, Log Rank; Hazard Ratio (HR) = 0.706, 95% CI 2-sided [0.501 to 0.994] — The hazard ratio and its 95% CI were based on Cox Regression Model, stratified by Prostate-specific antigen doubling time (PSADT) (≤ 6 months vs. > 6 months) and use of osteoclast-targeted therapy (No, Yes)

3. Secondary Outcome: Time to Pain Progression - Primary Analysis
Description: Time to pain progression (PP) is defined as time from randomization to pain progression, where progression is defined as an increase of 2 or more points from baseline in question 3 of the Brief Pain Inventory-Short Form questionnaire (BPI-SF) related to the worst pain in the last 24 hours taken as a 7-day average for post-baseline scores, or initiation of short or long-acting opioids for pain, whichever comes first. Initiation or change in the use of other non-opioid analgesics is not used in the analysis of pain progression.
Time Frame: From randomization until last study treatment (assessed every 4 months) (approximately 48 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Darolutamide (BAY1841788) | Placebo
Number analyzed (Participants) | 955 | 554
months | 40.31 [33.21 to 41.20] | 25.36 [19.09 to 29.63]
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) vs Placebo; Test type: Superiority; p = 0.000008, Log Rank; Hazard Ratio (HR) = 0.647, 95% CI 2-sided [0.533 to 0.785] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Time to Initiation of First Cytotoxic Chemotherapy for Prostate Cancer - Primary Analysis
Description: The time to cytotoxic chemotherapy was defined as the time from randomization to the start of the first cytotoxic chemotherapy cycle.
Time Frame: From randomization until last study treatment (assessed every 4 months) (approximately 48 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Darolutamide (BAY1841788) | Placebo
Number analyzed (Participants) | 955 | 554
months | NA [NA to NA] — NA = value cannot be estimated due to censored data, insufficient number of participants with events | 38.21 [35.55 to 41.89]
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) vs Placebo; Test type: Superiority; p < 0.000001, Log Rank; Hazard Ratio (HR) = 0.433, 95% CI 2-sided [0.314 to 0.595] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Time to First Symptomatic Skeletal Event (SSE) - Primary Analysis
Description: The time to the first SSE was defined as the time from randomization to the occurrence of the first SSE.
Time Frame: From randomization until last study treatment (assessed every 4 months) (approximately 48 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Darolutamide (BAY1841788) | Placebo
Number analyzed (Participants) | 955 | 554
months | NA [NA to NA] — NA = value cannot be estimated due to censored data, insufficient number of participants with events | NA [NA to NA] — NA = value cannot be estimated due to censored data, insufficient number of participants with events
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) vs Placebo; Test type: Superiority; p = 0.011262, Log Rank; Hazard Ratio (HR) = 0.428, 95% CI 2-sided [0.218 to 0.842] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Overall Survival - Final Analysis
Description: Overall Survival (OS) was defined as the time from randomization to death due to any cause. The final analysis was done at the time of the data cut-off (15 NOV 2019).
Time Frame: From randomization of the first subject to the time approximatively 254 death events were observed (approximately 56 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Darolutamide (BAY1841788) | Placebo
Number analyzed (Participants) | 955 | 554
months | NA [56.14 to NA] — NA = value cannot be estimated due to censored data, insufficient number of participants with events | NA [46.91 to NA] — NA = value cannot be estimated due to censored data, insufficient number of participants with events
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) vs Placebo; Test type: Superiority; p = 0.003048, Log Rank; Hazard Ratio (HR) = 0.685, 95% CI 2-sided [0.533 to 0.881] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Time to Pain Progression - Final Analysis
Description: For time to pain progression, the analysis performed using the primary completion cut-off data (03 SEP 2018) was considered final and no new analysis was performed for time to pain progression.
Time Frame: From randomization until last study treatment (assessed every 4 months) (approximately 48 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Darolutamide (BAY1841788) | Placebo
Number analyzed (Participants) | 955 | 554
months | 40.31 [33.21 to 41.20] | 25.36 [19.09 to 29.63]
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) vs Placebo; Test type: Superiority; p = 0.000008, Log Rank; Hazard Ratio (HR) = 0.647, 95% CI 2-sided [0.533 to 0.785] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Time to Initiation of First Cytotoxic Chemotherapy for Prostate Cancer - Final Analysis
Description: The time to cytotoxic chemotherapy was defined as the time from randomization to the start of the first cytotoxic chemotherapy cycle. The final analysis was done at the time of the data cut-off (15 NOV 2019).
Time Frame: From randomization until initiation of first cytotoxic chemotherapy treatment (approximately 59 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Darolutamide (BAY1841788) | Placebo
Number analyzed (Participants) | 955 | 554
months | NA [NA to NA] — NA = value cannot be estimated due to censored data, insufficient number of participants with events | NA [NA to NA] — NA = value cannot be estimated due to censored data, insufficient number of participants with events
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) vs Placebo; Test type: Superiority; p = 0.000044, Log Rank; Hazard Ratio (HR) = 0.579, 95% CI 2-sided [0.444 to 0.755] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Time to First Symptomatic Skeletal Event (SSE) - Final Analysis
Description: The time to the first SSE was defined as the time from randomization to the occurrence of the first SSE. The final analysis was done at the time of the data cut-off (15 NOV 2019).
Time Frame: From randomization until occurrence of first SSE event (approximately 59 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Darolutamide (BAY1841788) | Placebo
Number analyzed (Participants) | 955 | 554
months | NA [NA to NA] — NA = value cannot be estimated due to censored data, insufficient number of participants with events | NA [NA to NA] — NA = value cannot be estimated due to censored data, insufficient number of participants with events
Statistical Analysis 1: Comparison: Darolutamide (BAY1841788) vs Placebo; Test type: Superiority; p = 0.005294, Log Rank; Hazard Ratio (HR) = 0.484, 95% CI 2-sided [0.287 to 0.815] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 30 days after last treatment (last cut-off date 14 JUN 2021)
Groups:
- Darolutamide (DB): Participants received Darolutamide 600 mg (2 tablets of 300 mg) twice daily with food, equivalent to a total daily dose of 1200 mg (double blind [DB]).
- Darolutamide (DB+OL): Participants received Darolutamide 600 mg (2 tablets of 300 mg) twice daily with food, equal to a total daily dose of 1200 mg. Participants in the darolutamide treatment arm were ongoing with open-label darolutamide treatment (darolutamide double-blind [DB] + open-label [OL]).
- Placebo (DB): Participants received matching placebo 2 tablets twice daily with food (double blind [DB]).
- Placebo+Darolutamide (CO): Participants received matching placebo 2 tablets twice daily with food. Participants from the placebo arm crossed over to receive open-label darolutamide treatment (placebo-darolutamide cross-over [CO]).
Arm/Group | Darolutamide (DB) | Darolutamide (DB+OL) | Placebo (DB) | Placebo+Darolutamide (CO)
All-Cause Mortality (participants affected / at risk) | 155/954 | 224/954 | 137/554 | 16/170
Serious Adverse Events (participants affected / at risk) | 251/954 | 367/954 | 121/554 | 43/170
Other Adverse Events (participants affected / at risk) | 673/954 | 742/954 | 354/554 | 110/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darolutamide (DB) (N=954) | Darolutamide (DB+OL) (N=954) | Placebo (DB) (N=554) | Placebo+Darolutamide (CO) (N=170)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 8 (9) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 6 (6) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 4 (5) | 4 (5) | 2 (2) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 8 (11) | 9 (12) | 3 (3) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 8 (9) | 12 (14) | 4 (5) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (3) | 4 (5) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 11 (12) | 2 (3) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 3 (4) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Retinal vascular disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 3 (5) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plicated tongue (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Rectal stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (6) | 2 (3) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Death (General disorders) | 4 (4) | 6 (6) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 5 (7) | 7 (11) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perinephric abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 15 (18) | 20 (24) | 6 (6) | 1 (2)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 2 (3) | 3 (4) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (2) | 2 (3) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tick-borne viral encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 12 (13) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 2 (3) | 4 (10) | 0 (0) | 1 (1)
Acute endocarditis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Wound abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Severe acute respiratory syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Medical device site joint infection (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 4 (7) | 0 (0) | 1 (1)
Diverticulitis intestinal perforated (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (3) | 4 (5) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stenosis of vesicourethral anastomosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Heart injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flatback syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Incarcerated parastomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Biopsy prostate (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angiocardiogram (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 3 (4) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 4 (5) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 3 (4) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (3) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bulbar palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 2 (3) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 6 (6) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 4 (4) | 1 (2) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Perineurial cyst (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
IIIrd nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 5 (6) | 5 (6) | 2 (2) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (2) | 1 (3) | 0 (0) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 11 (13) | 25 (29) | 7 (7) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 8 (10) | 4 (4) | 2 (3)
Nephritis (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 4 (4) | 4 (4) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 16 (17) | 33 (37) | 20 (20) | 6 (6)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 7 (9) | 11 (13) | 3 (3) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 7 (7) | 3 (3) | 1 (1)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Prostate induration (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3) | 3 (5) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (6) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7) | 1 (1) | 1 (1)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder catheterisation (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orchidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nephrostomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Artificial urinary sphincter implant (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiotherapy to brain (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary resection (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Aortic thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 2 (2) | 2 (2) | 1 (2) | 0 (0)
Device occlusion (Product Issues) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darolutamide (DB) (N=954) | Darolutamide (DB+OL) (N=954) | Placebo (DB) (N=554) | Placebo+Darolutamide (CO) (N=170)
Anaemia (Blood and lymphatic system disorders) | 60 (76) | 93 (136) | 28 (33) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 13 (17) | 21 (27) | 4 (4) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 19 (20) | 26 (30) | 6 (8) | 3 (4)
Cataract (Eye disorders) | 11 (11) | 15 (16) | 5 (6) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 25 (27) | 35 (39) | 12 (14) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 14 (16) | 16 (19) | 14 (15) | 3 (3)
Constipation (Gastrointestinal disorders) | 65 (70) | 84 (94) | 36 (41) | 8 (11)
Diarrhoea (Gastrointestinal disorders) | 69 (87) | 87 (114) | 33 (37) | 15 (16)
Nausea (Gastrointestinal disorders) | 53 (59) | 60 (76) | 32 (37) | 6 (6)
Vomiting (Gastrointestinal disorders) | 17 (19) | 21 (24) | 10 (12) | 3 (3)
Asthenia (General disorders) | 37 (42) | 43 (53) | 20 (23) | 7 (8)
Fatigue (General disorders) | 126 (164) | 142 (198) | 47 (60) | 9 (9)
Oedema peripheral (General disorders) | 43 (49) | 57 (67) | 17 (19) | 4 (4)
Pyrexia (General disorders) | 18 (25) | 21 (28) | 5 (7) | 5 (9)
Bronchitis (Infections and infestations) | 13 (17) | 23 (30) | 9 (10) | 3 (3)
Influenza (Infections and infestations) | 28 (33) | 36 (42) | 8 (8) | 2 (2)
Nasopharyngitis (Infections and infestations) | 39 (50) | 56 (78) | 23 (27) | 8 (11)
Pneumonia (Infections and infestations) | 10 (11) | 22 (24) | 5 (5) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 26 (29) | 34 (40) | 10 (13) | 3 (7)
Urinary tract infection (Infections and infestations) | 44 (59) | 73 (130) | 31 (37) | 12 (12)
COVID-19 (Infections and infestations) | 0 (0) | 6 (6) | 0 (0) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 41 (44) | 62 (69) | 23 (27) | 7 (8)
Rib fracture (Injury, poisoning and procedural complications) | 16 (17) | 28 (30) | 8 (10) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 12 (17) | 21 (26) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 6 (8) | 13 (16) | 1 (1) | 6 (9)
Aspartate aminotransferase increased (Investigations) | 12 (16) | 23 (29) | 1 (1) | 6 (10)
Blood creatinine increased (Investigations) | 23 (32) | 37 (51) | 14 (19) | 3 (3)
Weight decreased (Investigations) | 40 (42) | 65 (72) | 14 (17) | 8 (8)
Weight increased (Investigations) | 14 (15) | 25 (27) | 7 (8) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 16 (24) | 22 (32) | 9 (10) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (10) | 12 (13) | 2 (2) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 30 (34) | 40 (49) | 16 (18) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 106 (146) | 135 (190) | 58 (69) | 17 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 92 (104) | 118 (142) | 52 (59) | 9 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 (20) | 20 (21) | 4 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (21) | 24 (28) | 7 (8) | 2 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 (20) | 26 (33) | 3 (3) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 60 (79) | 71 (105) | 19 (25) | 5 (6)
Dizziness (Nervous system disorders) | 39 (47) | 48 (64) | 14 (17) | 2 (2)
Headache (Nervous system disorders) | 41 (59) | 53 (75) | 14 (15) | 4 (7)
Depression (Psychiatric disorders) | 20 (20) | 25 (27) | 9 (10) | 2 (2)
Insomnia (Psychiatric disorders) | 26 (28) | 35 (38) | 11 (11) | 8 (8)
Dysuria (Renal and urinary disorders) | 24 (27) | 32 (37) | 27 (30) | 5 (5)
Haematuria (Renal and urinary disorders) | 37 (48) | 66 (96) | 27 (39) | 12 (13)
Nephrolithiasis (Renal and urinary disorders) | 14 (17) | 21 (25) | 4 (4) | 3 (3)
Nocturia (Renal and urinary disorders) | 17 (17) | 23 (24) | 10 (10) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 41 (46) | 51 (63) | 18 (20) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 15 (15) | 24 (25) | 14 (14) | 3 (3)
Urinary retention (Renal and urinary disorders) | 25 (27) | 39 (47) | 24 (29) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 21 (21) | 30 (30) | 6 (6) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 13 (15) | 16 (19) | 12 (13) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (34) | 33 (38) | 11 (11) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 (28) | 32 (34) | 16 (22) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (20) | 22 (25) | 12 (14) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 17 (17) | 24 (27) | 4 (4) | 2 (2)
Hypertension (Vascular disorders) | 66 (86) | 87 (117) | 31 (39) | 6 (7)
Hot flush (Vascular disorders) | 54 (58) | 67 (73) | 25 (25) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-07-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT02200614/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT02200614/SAP_003.pdf